CLINICAL TRIAL: NCT02621606
Title: A Three-Part Trial to Qualify [11C]MK-6884 Positron Emission Tomography for Use as a Biomarker for Regional M4 PAM Receptor Density Quantification in the Human Brain
Brief Title: [11C]MK-6884 Positron Emission Tomography (PET) Tracer Validation Trial (MK-6884-001)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 6884-001; MK-6884-001 (Other: Merck Protocol Number); 2015-001631-20 (EudraCT Number)
Record Dates: First submitted 2015-11-20; First posted 2015-12-03 (Estimated); Results first posted 2019-02-28 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-08

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part 1, Healthy Participants (Experimental): Healthy participants receive a single intravenous (IV) dose of ~370 megabecquerel (MBq) [11C]MK-6884 in Part 1 of the study.
  Interventions: Drug: [11C]MK-6884
- Part 2, Healthy Elderly Participants (Experimental): Healthy elderly participants receive two separate IV doses of ~370 MBq [11C]MK-6884 in Part 2 of the study. Administration of the two doses is separated by at least 3 hours.
  Interventions: Drug: [11C]MK-6884
- Part 3, Participants with AD (Experimental): Participants with AD receive a single IV dose of ~370 MBq [11C]MK-6884 in Part 3 of the study.
  Interventions: Drug: [11C]MK-6884

INTERVENTIONS:
Drug: [11C]MK-6884 — IV bolus dose of ~370 MBq [11C]MK-6884

SUMMARY:
The purpose of this open-label, 3-part study is to investigate the safety and efficacy of [11C]MK-6884 as a positron emission tomography (PET) imaging agent for quantifying muscarinic 4 (M4) positive allosteric modulator (PAM) receptor density in brain regions of interest. The study will enroll healthy participants (Parts 1 and 2) and participants with Alzheimer's Disease (AD) (Part 3). The primary efficacy hypothesis is that the average intra-subject test-retest (T-RT) variability of tracer uptake in brain regions of interest is ≤20%.

ELIGIBILITY:
Inclusion Criteria:

Part 1, 2 and 3:

* Male, or non-pregnant and non-breast feeding female of 18 to 55 years of age (Part 1) or 55 to 85 years of age (Parts 2 and 3); in addition:

  * Male participant who is sexually active with females of childbearing potential must be willing to use a condom from the first dose of study drug until 3 months post the last dose of study drug
  * Female participant with reproductive potential must have serum β-human chorionic gonadotropin (β-hCG) test result consistent with non-pregnant state at screening and agree to use two acceptable methods of birth control beginning at screening visit, during study and until 2 weeks after the last dose of study drug
  * Female participant of non-childbearing potential must be post-menopausal female (participant has been without menses for at least 1 year and has a follicle stimulating hormone [FSH] level in the postmenopausal range at screening), or surgically sterile female (status post hysterectomy, oophorectomy, or tubal ligation)
* Body Mass Index (BMI) ≤35 kg/m^2, with height ≤195 cm and weight ≤136 kg
* In good health (Part 1) or generally healthy (Parts 2 and 3) based on medical history, physical examination, vital sign measurements and electrocardiogram (ECG)
* Nonsmoker and/or has not used nicotine or nicotine-containing products for at least approximately 3 months

Part 2 Only:

* Willing to allow placement of an arterial catheter in the radial artery
* Mini Mental Status Examination (MMSE) score ≥27
* No history of subjective memory or other cognitive complaints
* No objective evidence of memory or cognitive impairment

Part 3 Only:

* Moderate to severe AD as defined by:

  * MMSE score ≤20
  * Meets National Institute of Neurological and Communicative Diseases and Stroke/Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria for probable AD
  * Meets Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-V) criteria for AD
  * Rosen-Modified Hachinski score ≤4
  * Screening magnetic resonance imaging (MRI) scan consistent with a diagnosis of AD
* Clear history of cognitive and functional decline over ≥1 year
* On a stable dose of one of protocol-defined acetylcholinesterase inhibitors (AChEIs) (i.e., donepezil and rivastigmine) for symptomatic treatment of AD. Dose must be stable for at least the last 4 weeks before screening
* Has a reliable trial partner/caregiver who is able to accompany the participant to all clinic visits, if needed, and able to provide information to study investigator/staff via telephone contact

Exclusion Criteria:

Part 1, 2, and 3:

* Mentally or legally incapacitated, has significant emotional problems at the time of screening visit or expected during the conduct of the trial or has a history of clinically significant psychiatric disorder of the last 5 years, except (for Part 3 only) for psychiatric disorders associated with AD
* History of clinically significant endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary or major neurological abnormalities or diseases, unless (for Part 2 and 3 only) adequately controlled through a stable medication regimen
* History of cancer
* History of significant multiple and/or severe allergies or has had an anaphylactic reaction or significant intolerability to prescription or non-prescription drugs or food. For Part 2, this includes any known allergy to lidocaine which may be used as an anesthetic for the placement of the arterial catheter
* Has positive test result for hepatitis B surface antigen, hepatitis C antibodies or human immunodeficiency virus (HIV)
* Has had major surgery or donated or lost 1 unit of blood (approximately 500 mL) within 4 weeks prior to screening
* Has participated in another investigational trial within 4 weeks of screening
* Corrected QT (QTc) interval ≥470 msec (for males) or ≥480 msec (for females)
* Is unable to refrain from or anticipates the use of any medication, including prescription and non-prescription drugs or herbal remedies, beginning approximately 2 weeks prior to administration of the initial dose of study drug and throughout the study.
* Consumes >3 servings of alcohol a day
* Consumes >6 caffeine servings a day
* Is currently a regular or recreational user of cannabis, any illicit drugs or has a history of drug (including alcohol) abuse within approximately 3 months
* Has participated in a PET research study or other study involving administration of a radioactive substance or ionizing radiation within 12 months prior to screening or has undergone an extensive radiological examination within this period
* Suffers from claustrophobia or an inability to tolerate confinement in small places and would be unable to undergo MRI or PET scanning

Part 2 Only:

- Has been administered an AChEI within the prior 3 months or will require administration of an AChEI during study

Part 3 Only:

* Has been administered galantamine within the prior 7 days or will require administration of galantamine during study
* History within 2 years prior to screening, or current evidence of any neurological or neurodegenerative disorder other than AD that is associated with transient or sustained alterations in cognition
* History within 2 years prior to screening, or current evidence of a psychotic disorder or a major depressive disorder

Part 2 and 3 Only:

- Has or is suspected to have implanted or embedded metal objects, or fragments in the head or body that would present a risk during the MRI scanning procedure

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-01-08 (Actual); Primary Completion 2017-12-28 (Actual); Study Completion 2017-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Li W, Wang Y, Lohith TG, Zeng Z, Tong L, Mazzola R, Riffel K, Miller P, Purcell M, Holahan M, Haley H, Gantert L, Hesk D, Ren S, Morrow J, Uslaner J, Struyk A, Wai JM, Rudd MT, Tellers DM, McAvoy T, Bormans G, Koole M, Van Laere K, Serdons K, de Hoon J, Declercq R, De Lepeleire I, Pascual MB, Zanotti-Fregonara P, Yu M, Arbones V, Masdeu JC, Cheng A, Hussain A, Bueters T, Anderson MS, Hostetler ED, Basile AS. The PET tracer [11C]MK-6884 quantifies M4 muscarinic receptor in rhesus monkeys and patients with Alzheimer's disease. Sci Transl Med. 2022 Jan 12;14(627):eabg3684. doi: 10.1126/scitranslmed.abg3684. Epub 2022 Jan 12. PMID 35020407

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy participants (Part 1), healthy elderly participants (Part 2), and participants with Alzheimer's Disease (AD; Part 3) were enrolled in this study.
Pre-assignment Details: N=20 participants were enrolled, with N=20 receiving ≥1 dose of [11C]MK-6884. N=1 participant in Part 2 withdrew from study before receiving the second dose of [11C]MK-6884.
Period: Overall Study
Arm/Group | Part 1, Healthy Participants | Part 2, Healthy Elderly Participants | Part 3, Participants With AD
Started | 3 | 7 | 10
Treated | 3 | 7 | 10
Completed | 3 | 6 | 10
Not Completed | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis population includes all randomized participants.
Groups:
- Part 1, Healthy Participants: Healthy participants receive a single IV dose of ~370 MBq [11C]MK-6884 in Part 1 of the study.
- Total: Total of all reporting groups
Arm/Group | Part 1, Healthy Participants | Part 2, Healthy Elderly Participants | Part 3, Participants With AD | Total
Number analyzed (Participants) | 3 | 7 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: Years] | 25.3 (2.1) | 62.6 (5.4) | 67.6 (5.2) | 59.5 (15.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 5 | 8
  Male | 2 | 5 | 5 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 3 | 7 | 9 | 19
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing an Adverse Event (AE)
Description: The number of participants experiencing an adverse event (AE) was assessed. An AE is defined as any unfavorable and unintended medical occurrence, sign, symptom, or disease temporally associated with the use of a pharmaceutical product or protocol-specified procedure, whether or not considered related to the pharmaceutical product or protocol-specified procedure. Any worsening of a preexisting condition, temporally associated with the use of the Sponsor's product, is also an AE.
Time Frame: Up to 15 days
Population: Includes all participants receiving ≥1 dose of [11C]MK-6884 in Parts 1, 2, or 3.
Measure: Count of Participants; unit: Participants
Groups:
- Part 1, Healthy Participants: Healthy participants receive a single IV dose of ~370 megabecquerel MBq [11C]MK-6884 in Part 1 of the study.
Arm/Group | Part 1, Healthy Participants | Part 2, Healthy Elderly Participants | Part 3, Participants With AD
Number analyzed (Participants) | 3 | 7 | 10
Participants | 1 | 5 | 1

2. Primary Outcome: Number of Participants Discontinuing the Study Due to an Adverse Event (AE)
Description: The number of participants discontinuing the study due to an AE was assessed. An AE is defined as any unfavorable and unintended medical occurrence, sign, symptom, or disease temporally associated with the use of a pharmaceutical product or protocol-specified procedure, whether or not considered related to the pharmaceutical product or protocol-specified procedure. Any worsening of a preexisting condition, temporally associated with the use of the Sponsor's product, is also an AE.
Time Frame: Up to 15 days
Population: Includes all participants receiving ≥1 dose of [11C]MK-6884 in Parts 1, 2, or 3.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1, Healthy Participants | Part 2, Healthy Elderly Participants | Part 3, Participants With AD
Number analyzed (Participants) | 3 | 7 | 10
Participants | 0 | 0 | 0

3. Primary Outcome: [Part 1] Mean Effective Dose of [11C]MK-6884
Description: Mean effective dose (ED) of [11C]MK-6884 was calculated as a measure of risk associated with exposure of the whole body (WB) to low levels of ionizing radiation. Following [11C]MK-6884 injection, WB positron emission tomography (PET) scans were collected to visually identify organs absorbing [11C]MK-6884 in significant amounts. Around identified organs, three-dimensional (3D) volumes were drawn to estimate the percentage of injected activity absorbed. These data were converted into time-activity curves (TACs) and retention of radioactivity in these regions was entered into a human biodistribution model to determine ED of [11C]MK-6884. ED is expressed in units millisieverts (mSv) / MBq.
Time Frame: Up to 2 hours post-dose
Population: Includes only healthy participants in Part 1 (N=3). Per protocol, participants in Parts 2 and 3 were not tested for ED of [11C]MK-6884 and are excluded.
Measure: Mean (Standard Deviation); unit: mSv / MBq
Arm/Group | Part 1, Healthy Participants | Part 2, Healthy Elderly Participants | Part 3, Participants With AD
Number analyzed (Participants) | 3 | 0 | 0
mSv / MBq | 0.0072 (0.00127) |  |

4. Primary Outcome: [Part 1] Mean Organ Effective Dose of [11C]MK-6884
Description: Mean organ ED of [11C]MK-6884 was calculated as a measure of risk associated with exposure of individual organs to low levels of ionizing radiation. Following [11C]MK-6884 injection, WB PET scans were collected to visually identify organs absorbing [11C]MK-6884 in significant amounts. Around identified organs, 3D volumes were drawn to estimate the percentage of injected activity absorbed. These data were converted into TACs and retention of radioactivity in these regions was used to calculate organ-specific ED of [11C]MK-6884. For sex organs (testes/ovaries), organ EDs were derived for participants of the respective sex. However, organ ED for the uterus was estimable in all participants as the male radiologic phantom was sufficiently hermaphroditic.
Time Frame: Up to 2 hours post dose
Population: Includes only healthy participants in Part 1 (N=3), having estimable data for the individual organ. Per protocol, participants in Parts 2 and 3 were not tested for organ ED of [11C]MK-6884 and are excluded.
Measure: Mean (Standard Deviation); unit: mSv / MBq
Arm/Group | Part 1, Healthy Participants | Part 2, Healthy Elderly Participants | Part 3, Participants With AD
Number analyzed (Participants) | 3 | 0 | 0
mSv / MBq
  Adrenals | 0.00000924 (0.0000019) |  |
  Brain | 0.00000666 (0.00000135) |  |
  Breasts | 0.0000804 (0.0000212) |  |
  Gallbladder Wall | 0 (0) |  |
  Lower Large Intestine Wall | 0.000499 (0.000146) |  |
  Small Intestine | 0.000802 (0.000217) |  |
  Stomach Wall | 0.000357 (0.0000962) |  |
  Upper Large Intestine Wall | 0.0000312 (0.00000782) |  |
  Heart Wall | 0 (0) |  |
  Kidneys | 0.0000476 (0.00000571) |  |
  Liver | 0.00104 (0.000236) |  |
  Lungs | 0.000709 (0.000228) |  |
  Muscle | 0.00000541 (0.00000144) |  |
  Ovaries (Female Participants Only): number analyzed (Participants) | 1 | 0 | 0
  Ovaries (Female Participants Only) | 0.00126 (0) |  |
  Pancreas | 0.00000938 (0.00000215) |  |
  Red Marrow | 0.000541 (0.0000553) |  |
  Osteogenic Cells | 0.000041 (0.0000106) |  |
  Skin | 0.0000145 (0.00000409) |  |
  Spleen | 0.0000256 (0.0000202) |  |
  Testes (Male Participants Only): number analyzed (Participants) | 2 | 0 | 0
  Testes (Male Participants Only) | 0.0017 (0.000573) |  |
  Thymus | 0.00000463 (0.00000118) |  |
  Thyroid | 0.0000732 (0.0000218) |  |
  Urinary Bladder Wall | 0.00135 (0.00045) |  |
  Uterus | 0.0000124 (0.00000334) |  |

5. Primary Outcome: [Part 2] Mean Non-displaceable Binding Potential (BPND) of [11C]MK-6884 in Brain Regions of Interest (ROI)
Description: Mean BPND of [11C]MK-6884 in each brain ROI was assessed. BPND is the ratio at equilibrium of specifically bound [11C]MK-6884 to that of non-displaceable [11C]MK-6884 in tissue. At time "0", a single IV bolus of [11]MK-6884 is administered and PET scanning initiated, yielding brain regional TACs. These TACs are then used to determine peak standard uptake value (SUV) and area under the curve (AUC) in order to quantify brain regional [11C]MK-6884 uptake. The target region BPND is estimated using the cerebellum as the reference region with the transient equilibrium tissue ratio (TE-TR) method. Higher values indicate increased specific [11C]MK-6884 binding in the brain ROI.
Time Frame: Up to 90 minutes post dose
Population: Includes only healthy elderly participants in Part 2 receiving 2 doses of [11C]MK-6884 who sufficiently comply with study protocol (N=6). Per protocol, participants in Part 1 were not tested for mean BPND of [11C]MK-6884 and are excluded. Mean BPND data for Part 3 participants are presented in a separate table.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Part 1, Healthy Participants | Part 2, Healthy Elderly Participants | Part 3, Participants With AD
Number analyzed (Participants) | 0 | 6 | 0
Ratio
  Putamen |  | 1.15 (0.14) |
  Striatum |  | 0.96 (0.13) |
  Frontal Cortex |  | 0.92 (0.15) |
  Temporal Cortex |  | 0.92 (0.12) |
  Hippocampus |  | 0.45 (0.11) |

6. Primary Outcome: [Part 2] Intra-subject Test-Retest (T-RT) Variability of Non-displaceable Binding Potential (BPND) of [11C]MK-6884 in Brain Regions of Interest (ROI)
Description: Intra-subject T-RT variability in BPND of [11C]MK-6884 in each brain ROI was assessed. For each healthy elderly participant receiving 2 doses of [11C]MK-6884 in study Part 2, the BPND calculated during the first dose (BPND-1) was compared to the BPND calculated during the second dose (BPND-2) to determine the percent T-RT variability of the BPND of [11C]MK-6884 for each brain ROI.
  Percent T-RT variability = [absolute value (BPND-1 - BPND-2) / (average BPND)] * 100. A percent T-RT variability = 0, indicates no variability between BPND-1 and BPND-2.
Time Frame: Up to 24 hours post dose
Population: Includes only healthy elderly participants in Part 2 receiving 2 doses of [11C]MK-6884 who sufficiently comply with study protocol (N=6). Per protocol, participants in Parts 1 and 3 were not tested for intra-subject T-RT variability of BPND of [11C]MK-6884 and are excluded.
Measure: Mean (Standard Deviation); unit: Percent variability
Arm/Group | Part 1, Healthy Participants | Part 2, Healthy Elderly Participants | Part 3, Participants With AD
Number analyzed (Participants) | 0 | 6 | 0
Percent variability
  Putamen |  | 14.1 (9.0) |
  Striatum |  | 11.1 (9.2) |
  Frontal Cortex |  | 16.0 (7.8) |
  Temporal Cortex |  | 10.9 (13.7) |
  Hippocampus |  | 24.9 (15.3) |

7. Primary Outcome: [Part 3] Mean Regional Non-displaceable Binding Potential (BPND) of [11C]MK-6884 in Brain Regions of Interest
Description: Mean BPND of [11C]MK-6884 in each brain ROI was assessed. BPND is the ratio at equilibrium of specifically bound [11C]MK-6884 to that of non-displaceable [11C]MK-6884 in tissue. At time "0", a single IV bolus of [11]MK-6884 is administered and PET scanning initiated, yielding brain regional TACs. These TACs are then used to determine SUV and AUC in order to quantify brain regional [11C]MK-6884 uptake. The target region BPND is estimated using the cerebellum as the reference region with the TE-TR method. Higher values indicate increased specific [11C]MK-6884 binding in the brain ROI.
Time Frame: Up to 90 minutes post dose
Population: Includes only participants with AD in Part 3 receiving [11C]MK-6884 who sufficiently comply with study protocol (N=10). Per protocol, participants in Part 1 were not tested for mean BPND of [11C]MK-6884 and are excluded. Mean BPND data for Part 2 participants are presented in a separate table.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Part 1, Healthy Participants | Part 2, Healthy Elderly Participants | Part 3, Participants With AD
Number analyzed (Participants) | 0 | 0 | 10
Ratio
  Frontal Cortex |  |  | 0.74 (0.20)
  Striatum |  |  | 0.98 (0.20)

ADVERSE EVENTS:
Time Frame: Up to 15 days
Description: An AE is defined as any unfavorable and unintended medical occurrence, sign, symptom, or disease temporally associated with the use of a pharmaceutical product or protocol-specified procedure, whether or not considered related to the pharmaceutical product or protocol-specified procedure. Any worsening of a preexisting condition, temporally associated with the use of the Sponsor's product, is also an AE. All participants receiving ≥1 dose of [11C]MK-6884 in study Parts 1, 2, or 3 are included.
Arm/Group | Part 1, Healthy Participants | Part 2, Healthy Elderly Participants | Part 3, Participants With AD
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/7 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/7 | 0/10
Other Adverse Events (participants affected / at risk) | 1/3 | 4/7 | 1/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1, Healthy Participants (N=3) | Part 2, Healthy Elderly Participants (N=7) | Part 3, Participants With AD (N=10)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1, Healthy Participants (N=3) | Part 2, Healthy Elderly Participants (N=7) | Part 3, Participants With AD (N=10)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Glossodynia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Lip dry (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 0 (0)
Procedural nausea (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness postural (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-24): https://cdn.clinicaltrials.gov/large-docs/06/NCT02621606/Prot_SAP_000.pdf